CLINICAL TRIAL: NCT04836247
Title: Understanding and Addressing Disclosure to Members of Social Networks Among People Recovering From Substance Use Disorders
Brief Title: Disclosure Intervention for People in Recovery From Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Massachusetts General Hospital (Other); Harvard School of Public Health (HSPH) (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Valerie Earnshaw, Associate Professor of Human Development and Family Sciences, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K01DA042881 (NIH); K01DA042881 (NIH)
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Opioid-use Disorder
Keywords: disclosure; social support; stigma; patient decision aid
MeSH Terms: conditions — Opioid-Related Disorders; Social Stigma | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disclosure Intervention Arm (Experimental): Participants will be guided through a workbook and accompanying worksheet designed to help them: (1) decide whether or not they want to share information about their substance use with others, and (2) build skills for disclosing (e.g., planning what to say). Importantly, the intervention is not designed to encourage participants to disclose or not disclose, but rather to help participants decide whether they want to disclose based on their own goals and values.
  Interventions: Behavioral: Disclosing Recovery: A Decision Aid and Toolkit
- Control Arm (Active Comparator): Participants will be able to choose from several guided meditations to promote mindfulness.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Disclosing Recovery: A Decision Aid and Toolkit — Participants will be guided through a workbook and accompanying worksheet designed to help them: (1) decide whether or not they want to share information about their substance use with others, and (2) build skills for disclosing (e.g., planning what to say). Importantly, the intervention is not designed to encourage participants to disclose or not disclose, but rather to help participants decide whether they want to disclose based on their own goals and values.
  Arms: Disclosure Intervention Arm
Behavioral: Mindfulness — Participants will be able to choose from several guided meditations to promote mindfulness
  Arms: Control Arm

SUMMARY:
Many people with substance use disorders struggle with decisions regarding whether to disclose to others that they have a history of substance use and/or are in recovery. Yet, these decisions are important because disclosures can lead to reactions from others that harm or help recovery. For example, stigmatizing responses can harm the mental health of people in recovery whereas supportive responses can strengthen people's commitment to their sobriety. We have developed a brief intervention to help people decide whether and how to tell others about their recovery as well as build skills for disclosure. The purpose of this study is to pilot test this intervention and test its acceptability and feasibility as well as determine if it shows preliminary signs of efficacy in comparison to a control condition. We hypothesize that: (1) participants exposed to the intervention condition will agree that the intervention is acceptable and feasible, and (2) participants in the intervention condition will report higher quality decision making in comparison to participants in the control condition.

DETAILED DESCRIPTION:
Data will be collected from participants at two time points, spaced one month apart. All participants will be recruited from the waiting room at a local treatment center. The research assistant will screen interested individuals for eligibility in person and schedule study appointments, which may be coordinated with treatment appointments. All study screening and appointments will be conducted in private spaces at the treatment center. At the first study appointment, the research assistant will introduce the study, check for questions, and obtain consent for the study procedures, medical record review, and follow up procedures. Participants will be randomly assigned to receive either the disclosure intervention or a control intervention (i.e., an evidence-based mindfulness intervention). Following the intervention, participants will complete measures of acceptability, feasibility, and decision quality. At the second study appointment, participants will again be asked to respond to survey and interview questions designed to further evaluate the preliminary efficacy of the intervention. In particular, we will investigate whether participants who completed our disclosure intervention report better relationship outcomes than participants who completed the control condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* currently receiving outpatient treatment at the recruitment site
* are considering disclosing their recovery status to at least one person in the next month
* have access to a phone that can receive text messages and phone calls

Exclusion Criteria:

* current diagnosis of severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brandywine Counseling and Community Services, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Earnshaw VA, Sepucha KR, Laurenceau JP, Subramanian SV, Hill EC, Wallace J, Brousseau NM, Henderson C, Brohan E, Morrison LM, Kelly JF. Disclosing Recovery: A pilot randomized controlled trial of a patient decision aid to improve disclosure processes for people in treatment for opioid use disorder. J Subst Use Addict Treat. 2024 May;160:209291. doi: 10.1016/j.josat.2024.209291. Epub 2024 Jan 23. PMID 38272118

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Disclosure Intervention Arm | Control Arm
Started | 25 | 25
Completed | 25 (25 participants responded to primary outcome measures, 24-25 responded to secondary outcome measures) | 25 (25 participants responded to primary outcome measures, 24-25 responded to secondary outcome measures. 1 participant was excluded from secondary outcome analyses (due to missing data))
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disclosure Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.04 (10.94) | 42.04 (11.32) | 41.54 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 22 | 20 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention
Description: Measured with Acceptability of Intervention Measure (adapted from Weiner et al., 2017). Mean scores range 1-5, with higher scores indicating greater acceptability.
Time Frame: Assessed immediately following intervention delivery, at time 1 study appointment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Disclosure Intervention Arm | Control Arm
Number analyzed (Participants) | 25 | 25
score on a scale | 4.82 (0.34) | 3.19 (1.14)
Statistical Analysis 1: Comparison: Disclosure Intervention Arm vs Control Arm; Test type: Superiority; p < .001, t-test, 2 sided — <.001 is calculated p-value in SPSS; Mean Difference (Final Values) = 1.63

2. Primary Outcome: Feasibility of Intervention
Description: Measured with Feasibility of Intervention Measure (adapted from Weiner et al., 2017). Mean scores range 1-5, with higher scores indicating greater feasibility.
Time Frame: Assessed immediately following intervention delivery, at time 1 study appointment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Disclosure Intervention Arm | Control Arm
Number analyzed (Participants) | 25 | 25
score on a scale | 4.88 (0.32) | 3.78 (0.84)
Statistical Analysis 1: Comparison: Disclosure Intervention Arm vs Control Arm; Test type: Superiority; p < .001, t-test, 2 sided — <.001 is calculated p-value in SPSS; Mean Difference (Final Values) = 1.10

3. Primary Outcome: Decision Making Quality
Description: Measured informed by recommendations for evaluating patient decision aids (Sepucha et al., 2013), focused on recognition of decision. Mean scores range 1-5, with higher scores indicating greater decision making quality.
Time Frame: Assessed immediately following intervention delivery, at time 1 study appointment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Disclosure Intervention Arm | Control Arm
Number analyzed (Participants) | 25 | 25
score on a scale | 4.49 (0.59) | 1.88 (0.98)
Statistical Analysis 1: Comparison: Disclosure Intervention Arm vs Control Arm; Test type: Superiority; p < .001, t-test, 2 sided — <.001 is calculated p-value in SPSS; Mean Difference (Final Values) = 2.61

4. Secondary Outcome: Social Support
Description: Measure adapted from Medical Outcomes Study Social Support Survey (Moser et al., 2012); Mean scores range 1-5, higher scores indicate more social support.
Time Frame: Second study appointment out of two. Second appointment took place approximately one month after first study appointment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Disclosure Intervention Arm | Control Arm
Number analyzed (Participants) | 24 | 23
score on a scale | 3.17 (1.17) | 3.29 (1.38)
Statistical Analysis 1: Comparison: Disclosure Intervention Arm vs Control Arm; Test type: Superiority; p = 0.74, t-test, 2 sided; Mean Difference (Final Values) = -0.12

5. Secondary Outcome: Enacted Stigma
Description: Measure adapted from Methadone Maintenance Treatment Stigma Mechanisms Scale (Smith et al., 2019); Mean scores range 1-5, higher scores indicate greater stigma.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Disclosure Intervention Arm | Control Arm
Number analyzed (Participants) | 24 | 23
score on a scale | 1.83 (0.72) | 1.91 (1.03)
Statistical Analysis 1: Comparison: Disclosure Intervention Arm vs Control Arm; Test type: Superiority; p = 0.76, t-test, 2 sided; Mean Difference (Final Values) = -0.08

6. Secondary Outcome: Commitment to Sobriety
Description: Measured with Commitment to Sobriety Scale (Kelly & Greene, 2014); Mean scores range 1-6, higher scores indicate greater commitment to sobriety.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Disclosure Intervention Arm | Control Arm
Number analyzed (Participants) | 24 | 23
score on a scale | 5.48 (0.70) | 5.62 (0.53)
Statistical Analysis 1: Comparison: Disclosure Intervention Arm vs Control Arm; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = 0.14

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Disclosure Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04836247/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04836247/ICF_001.pdf